CLINICAL TRIAL: NCT05264740
Title: Motivational Interviewing to Promote Healthy Behaviours for Obesity Prevention in Young Adults: a Pilot Randomized Controlled Trial
Brief Title: Motivational Interviewing to Promote Healthy Behaviours in Young Adults
Acronym: Motivate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 707228
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Risk Factors
Keywords: prevention; young adult; exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental)
  Interventions: Behavioral: Motivational interviewing
- no motivational interviewing (Active Comparator)
  Interventions: Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Motivational interviewing — The intervention group will receive motivational interviewing sessions with a trained study nurse plus educational material
  Arms: Motivational interviewing
Behavioral: Educational materials — The control group will receive educational material only.
  Arms: no motivational interviewing

SUMMARY:
The overall goals of this project are to evaluate the feasibility of web-based nurse-led motivational interviewing and educational interventions to promote healthy behaviours for obesity prevention and maintenance of healthy weight and behaviours among young adults attending university (age 18-29) in Hamilton, Ontario. A secondary goal is to evaluate if the intervention is more successful among people at higher risk of obesity (a risk stratification approach). A pilot randomized controlled trial will be conducted. Young adults will be randomized to receive a tailored behavioural intervention through motivational interviewing sessions with a nurse combined with educational materials, or control (educational materials only). Both groups will be followed for 6 months and their weight at baseline and end of the study will be measured. Outcomes related to the feasibility of the intervention and participants' experiences in the study will also be measured.

DETAILED DESCRIPTION:
Obesity is an established risk factor for many cancer types, including colon, endometrial, breast, and pancreatic. Obesity is complex and treatment is challenging. Thus, primary prevention of obesity is important. This is particularly important now since the COVID-19 pandemic had a profound impact on many obesity risk factors, such as chronic stress, overeating, and physical inactivity. Early adulthood is a key period in obesity development and a critical period for prevention interventions. Young adulthood is a period when Canadians may be highly amenable to healthy behaviour change, develop lifelong healthy behaviours and the primary prevention of obesity may be feasible. Interventions in early adulthood have the potential for primordial cancer prevention (i.e., stopping cancer risk factors before they develop). Despite the known impact of obesity on cancer, there have been few attempts to implement tailored population-based obesity prevention interventions. Obesity interventions must be flexible to address the complex causes of obesity and motivational interviewing may be a successful strategy.

Primary Objective:

1. To determine the feasibility (enrollment, retention, data completion, satisfaction) of a 6-month behavioural and educational intervention to promote healthy behaviours for obesity prevention among young adults.

   Secondary objectives:
2. To determine the effects of the 6-month behavioural and educational intervention, compared to an educational intervention only, on change in BMI, health behaviours (nutrition, physical activity and sedentary time) and mental health (depression and anxiety)
3. To explore whether obesity risk stratification tools identify young adults who may be more successful in an obesity intervention.

Methods: A pilot randomized controlled trial will be conducted. Young adults (age 18-29) attending McMaster University will be recruited and randomized to either the intervention or control. The intervention will include individual motivational interviewing sessions (online or in-person) with a trained public health nurse plus educational materials (based on Canada's food guide and physical activity recommendations). The control group will receive educational materials only. The primary feasibility outcomes that will be evaluated as part of this pilot study include enrollment, retention (≥80%), data completion (≥80% of weights measured, and surveys completed), and participant satisfaction. Clinical outcomes will include weight change from baseline to 6-months, physical activity, nutrition risk, and mental health. Outcomes will be measured remotely using 'smart' electronic scales, activity trackers, and online questionnaires at baseline and every 2 months. Risk stratification will be applied at baseline to identify participants at high risk of obesity (e.g., due to family or personal history). Exit questionnaires will collect data on how participants felt about the study and cost analysis will be conducted.

Our proposed evaluation of the feasibility of an obesity prevention intervention in early adulthood will inform future larger RCTs for obesity prevention. The results of this study have the potential to directly contribute to the primary prevention of several types of cancer by testing an intervention that could be scalable to public health, post-secondary education, or primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, and capable of providing informed consent
* McMaster University students 18-29 years of age
* Body mass index of at least 18.5

Exclusion Criteria:

* Physical and mental health conditions that would be contraindicated for a weight management intervention, including eating disorders, pregnancy, cancer, or medications that affect body weight

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Anderson, PhD, Principal Investigator — McMaster University; Lawrence Mbuagbaw, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
For this pilot study, individual data will not be available.

REFERENCES:
- [Derived] Anderson LN, Alvarez E, Incze T, Tarride JE, Kwan M, Mbuagbaw L. Motivational interviewing to promote healthy behaviors for obesity prevention in young adults (MOTIVATE): a pilot randomized controlled trial protocol. Pilot Feasibility Stud. 2023 Sep 7;9(1):156. doi: 10.1186/s40814-023-01385-0. PMID 37679845

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interviewing: Motivational interviewing: The intervention group will receive motivational interviewing sessions with a trained study team member plus educational material
Period: Baseline
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Started | 52 | 49
Completed | 52 | 48
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow Up 1
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Started | 52 | 48
Completed | 51 | 46
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Follow Up 2
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Started | 51 | 46
Completed | 50 | 42
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 4
Period: Follow Up 3
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Started | 50 | 42
Completed | 43 | 38
Not Completed | 7 | 4
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Population: A total of 101 participants were randomized (52 to the Motivational Interviewing group, 49 to the No Motivational Interviewing group). One participant withdrew from the No Motivational Interviewing group before completing baseline characteristics, resulting in 100 participants. analyzed at baseline. For race/ethnicity participants were permitted to select "all that apply".
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing | no Motivational Interviewing | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.8 (3.49) | 23 (3.61) | 22.2 (3.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 28 | 26 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5 | 0 | 5
  East Asian | 10 | 9 | 19
  Southeast Asian | 0 | 2 | 2
  South Asian | 18 | 12 | 30
  Latino | 1 | 2 | 3
  Middle Eastern | 10 | 17 | 27
  White | 6 | 5 | 11
  Other | 0 | 2 | 2
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 24.6 (4.43) | 25.6 (5.27) | 25.1 (4.85)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: % of eligible participants who are recruited from all those who contact the research team to learn about the study
Time Frame: At recruitment, over 6 months.
Measure: Count of Participants; unit: Participants
Groups:
- Recruitment: All participants screened for eligibility.
Arm/Group | Recruitment
Number analyzed (Participants) | 118
Participants | 101

2. Primary Outcome: Retention Rate
Description: % of participants who complete 6-month follow-up
Time Frame: from 0 to 6 months
Measure: Number; unit: participants
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 52 | 49
participants | 43 | 38

3. Primary Outcome: Data Completion
Description: Number of participants with no missing data on clinical outcomes
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 52 | 49
Participants | 48 | 45

4. Primary Outcome: Study Satisfaction
Description: Satisfaction was measured using a single-item question:
  "How satisfied are you with this research study?"
  Responses were collected on a 5-point Likert scale with the following options:
  1. = Highly Dissatisfied
  2. = Dissatisfied
  3. = Neither Satisfied nor Dissatisfied
  4. = Satisfied
  5. = Highly Satisfied Mean scores were calculated, with higher scores indicating greater satisfaction.
Time Frame: At 6 months
Population: All participants who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 43 | 38
units on a scale | 3.8 (1.02) | 3.9 (1.05)

5. Secondary Outcome: Body Mass Index (BMI) Change
Description: Change in BMI from baseline to 6-month follow-up
Time Frame: Change from 0 to 6 months
Population: Discrepancy in Overall Number Analyzed due to missing data.
Measure: Mean (Standard Deviation); unit: kg/m²
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 46 | 42
kg/m² | -0.3 (0.89) | -0.5 (1.52)

6. Secondary Outcome: Physical Activity
Description: Minutes per day from activity trackers and International Physical Activity Questionnaire (IPAQ).Participants self-reported the number of days per week they engaged in moderate and vigorous physical activity using items adapted from the International Physical Activity Questionnaire (IPAQ). Responses ranged from 0 to 7 days per week for each activity type.
Time Frame: At 6 months
Population: Data from the IPAQ were available for 81 participants. Two participants in the control group had missing responses for the vigorous activity question, and two had missing responses for the moderate activity question. All participants in the intervention group completed both items.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 44 | 37
Participants
  Vigorous activity (0 days) | 14 | 12
  Vigorous activity (1-3 days) | 19 | 19
  Vigorous activity (4-6 days) | 11 | 6
  Vigorous activity (7 days) | 0 | 0

7. Secondary Outcome: Sedentary Time
Description: Measured per day from activity trackers and questionnaire. Sedentary behaviour was assessed using the International Sedentary Assessment Tool (ISAT).
Time Frame: At 6 months
Population: Data on sedentary behavior were available for 82 participants. One participant in the control group did not complete the ISAT, while all participants in the intervention group provided complete data.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 44 | 38
hours
  Sitting (pastime) (hrs) | 5 [3 to 7.4] | 4 [2.6 to 6]
  Driving (hrs) | 1 [0.5 to 2] | 1 [0.5 to 2]
  Sitting (full day) (hrs) | 7.9 [5 to 10] | 8 [6 to 9.9]

8. Secondary Outcome: Nutrition
Description: Measured from National Cancer Institute's Dietary Screener Questionnaire. Items from the National Cancer Institute's Dietary Screener Questionnaire (DSQ), which asked participants how often they consumed fruit over the past month. Responses ranged from "Never" to "More than once a day" and were reported separately for each item as frequency categories (n, %).
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 43 | 37
Participants
  <1 time per week | 6 | 7
  1-5 times/week | 25 | 20
  ≥1 time/day | 12 | 10

9. Secondary Outcome: Mental Health
Description: Depressive Symptoms- defined by the Center for Epidemiologic Studies Depression Scale (CES-D). >=10 indicating presence of depressive symptoms, <10 no depressive symptoms.
Time Frame: At 6 months
Population: Discrepancy in number analyzed due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | no Motivational Interviewing
Number analyzed (Participants) | 44 | 39
Participants
  Yes (>=10) | 23 | 20
  No (<10) | 21 | 19

ADVERSE EVENTS:
Time Frame: 6 months
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Motivational Interviewing | no Motivational Interviewing
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/52 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT05264740/Prot_SAP_000.pdf